CLINICAL TRIAL: NCT02407925
Title: Implementation of Optical Diagnosis for Diminutive Polyps Amongst Accredited Endoscopists for the Dutch Bowel Cancer Screening Program: Training and Long-term Quality Assurance
Brief Title: Implementation of Optical Diagnosis for Diminutive Polyps Amongst Endoscopists: Training and Long-term Quality Assurance
Acronym: DISCOUNT2
Status: Completed | Type: Observational
Sponsor: Academisch Medisch Centrum - Universiteit van Amsterdam (AMC-UvA) (Other)
Collaborators: Dutch Digestive Diseases Foundation (Other)
Responsible Party: Principal Investigator, Prof. Evelien Dekker, MD, PhD, MD, PhD, Academisch Medisch Centrum - Universiteit van Amsterdam (AMC-UvA)
Other Study IDs: W14_099; NTR4635 (Registry Identifier: The Netherlands National Trial Register); FP 13 (Other Grant/Funding Number: Dutch Digestive Foundation)
Record Dates: First submitted 2015-03-19; First posted 2015-04-03 (Estimated); Last update posted 2018-01-09 (Actual); Status verified 2018-01

CONDITIONS: Colonoscopy; Colonic Polyps
Keywords: Optical diagnosis
MeSH Terms: conditions — Colonic Polyps

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (3):
- Endoscopists: Approximately 35 endoscopists whom are certified to perform colonoscopies on FIT-positive patients in the Dutch population screening program
  Interventions: Behavioral: Feedback
- Colonoscopies: Colonoscopies on FIT-positive patients in the Dutch population screening program
- Device: Olympus colonoscopes with Narrow Band Imaging

INTERVENTIONS:
Behavioral: Feedback — 3-monthly or no 3-monthly feedback on results of optical diagnosis
  Groups: Endoscopists

SUMMARY:
In this study, Dutch gastroenterologists who are certified for performing colonoscopies on FIT-positive patients in the Dutch population screening program are trained in optical diagnosis with validated methods. After this training, an ex- and in-vivo test phase leads to "accreditation" and endoscopists will be observed in their optical diagnosis for 1 year. During this year, half of the endoscopists will be randomized towards 3-monthly feedback and the other half will receive feedback on their results after 1 year. The endoscopic prediction of endoscopists on polyp histology will be compared to histopathological outcome.

DETAILED DESCRIPTION:
Through the recently started nationwide bowel cancer screening programme in the Netherlands, an extra 70.000 colonoscopies are annually performed. In current practice, all resected colonic lesions are histopathologically analysed. Even diminutive polyps, which rarely harbour cancer or advanced histological features. If endoscopists are able to accurately differentiate between neoplastic and non-neoplastic lesions during colonoscopy, practice could become more efficient and costeffective. This strategy is called optical diagnosis and two clinical practice strategies have been proposed by the American Society of Gastroenterologists (ASGE). First, diminutive polyps could be resected and discarded if >90% of the surveillance intervals predicted on optical diagnosis correlate with the surveillance intervals after histopathological validation (if assessed with high confidence). Second, hyperplastic polyps in the rectosigmoid could be left in situ if endoscopists are able to confidently predict neoplastic histology of diminutive colorectal polyps with a negative predictive value (NPV) of ≥90%.

The accuracy of white light colonoscopy is not acceptable for daily practice (59%-84%), but narrow band imaging (NBI) allows higher accuracies up to 98% and it was demonstrated that experienced endoscopists could reach a NPV of ≥90% for diminutive colorectal lesions. However, recent research shows that community gastroenterologists are not able to meet the quality thresholds proposed by the ASGE. Before this strategy could be safely applied in daily practice, community gastroenterologists should be able to meet thresholds as well.

In this study, Dutch gastroenterologists who are certified for performing colonoscopies on FIT-positive patients in the Dutch population screening program, are trained in optical diagnosis with validated methods. After training, an ex- and in-vivo test phase leads to "accreditation" and endoscopists will be observed in their optical diagnosis for 1 year. During this year, half of the endoscopists will be randomized towards 3-monthly feedback and the other half will receive feedback on their results after 1 year. The endoscopic prediction of endoscopists on polyp histology will be compared to histopathological outcome.

ELIGIBILITY:
Inclusion Criteria:

* Colonoscopies performed in FIT positive patients obtained for the Dutch colorectal cancer screening program.

Exclusion Criteria:

* Colonoscopies in patients with a history of colorectal cancer, inflammatory bowel disease or polyposis syndrome.
* Colonoscopies in patients with bleeding disorders or anticoagulants and therefore cannot undergo polypectomy.

Ages: 55 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Endoscopists certified for performing Dutch screening colonoscopies. Colonoscopies in patients performed after a positive FIT obtained for the Dutch colorectal cancer screening program.
Sampling Method: Non-Probability Sample
Enrollment: 3144 (Actual)
Dates: Start 2015-01-01 (Actual); Primary Completion 2017-02-28 (Actual); Study Completion 2018-01-01 (Actual)

PRIMARY OUTCOMES:
the number of training rounds needed until endoscopists reach a clinical acceptable accuracy of predicting histology of subcentimetric (1-9 mm) colorectal lesions using NBI | 18 months
the number of qualified endoscopists that are able to maintain a clinical acceptable accuracy of predicting histology of subcentimetric (1-9 mm) colorectal lesions using NBI over a year, either with and without regular interim feedback. | 18 months

SECONDARY OUTCOMES:
the number of the accredited endoscopists that is able to reach a negative predictive value of at least 90% for predicting neoplastic diminutive (1-5mm) and small (6-9mm) colorectal lesions in the rectosigmoid | 18 months
the number of diminutive (1-5mm) and small (6-9mm) lesions that are correctly predicted with high confidence | 18 months
the number of patients in whom a surveillance interval (according to the Dutch surveillance guideline) can be advised directly after colonoscopy, based on the endoscopic diagnosis | 18 months
the number of patients in whom the surveillance interval (according to the Dutch surveillance guideline) is correctly predicted based on endoscopic diagnosis | 18 months
the number of correctly diagnosed sessile serrated adenoma/polyps in diminutive (1-5mm) and small (6-9mm) polyps | 18 months
the sensitivity for predicting neoplastic histology per endoscopist, time frame and feedback or no feedback group | 18 months
the costs in euros that would have been saved by multiplying the amount of high confidence predicted diminutive and small polyps with the histopathology costs per lesion | 18 months

CONTACTS AND LOCATIONS:
Overall Officials: Evelien Dekker, Prof. dr., Principal Investigator — e.dekker@amc.uva.nl
Locations (13):
- Netherlands (13):
  - Medisch Centrum Alkmaar, Alkmaar
  - Flevoziekenhuis, Almere Stad
  - Amstelland Ziekenhuis, Amstelveen
  - Antonie van Leeuwenhoek Ziekenhuis, Amsterdam
  - Onze Lieve Vrouwe Gasthuis, Amsterdam
  - Sint Lucas Andreas Ziekenhuis, Amsterdam
  - Slotervaart Ziekenhuis, Amsterdam
  - Rode Kruis Ziekenhuis, Beverwijk
  - Kennemer Gasthuis, Haarlem
  - Spaarne Ziekenhuis, Hoofddorp
  - West Fries Gasthuis, Hoorn
  - Sint Antonius Ziekenhuis, Nieuwegein
  - Diakonessenhuis, Utrecht

REFERENCES:
- [Background] Ignjatovic A, East JE, Suzuki N, Vance M, Guenther T, Saunders BP. Optical diagnosis of small colorectal polyps at routine colonoscopy (Detect InSpect ChAracterise Resect and Discard; DISCARD trial): a prospective cohort study. Lancet Oncol. 2009 Dec;10(12):1171-8. doi: 10.1016/S1470-2045(09)70329-8. Epub 2009 Nov 10. PMID 19910250
- [Background] Kuiper T, Marsman WA, Jansen JM, van Soest EJ, Haan YC, Bakker GJ, Fockens P, Dekker E. Accuracy for optical diagnosis of small colorectal polyps in nonacademic settings. Clin Gastroenterol Hepatol. 2012 Sep;10(9):1016-20; quiz e79. doi: 10.1016/j.cgh.2012.05.004. Epub 2012 May 18. PMID 22609999
- [Background] Rex DK, Kahi C, O'Brien M, Levin TR, Pohl H, Rastogi A, Burgart L, Imperiale T, Ladabaum U, Cohen J, Lieberman DA. The American Society for Gastrointestinal Endoscopy PIVI (Preservation and Incorporation of Valuable Endoscopic Innovations) on real-time endoscopic assessment of the histology of diminutive colorectal polyps. Gastrointest Endosc. 2011 Mar;73(3):419-22. doi: 10.1016/j.gie.2011.01.023. PMID 21353837
- [Background] Kaminski MF, Hassan C, Bisschops R, Pohl J, Pellise M, Dekker E, Ignjatovic-Wilson A, Hoffman A, Longcroft-Wheaton G, Heresbach D, Dumonceau JM, East JE. Advanced imaging for detection and differentiation of colorectal neoplasia: European Society of Gastrointestinal Endoscopy (ESGE) Guideline. Endoscopy. 2014 May;46(5):435-49. doi: 10.1055/s-0034-1365348. Epub 2014 Mar 17. PMID 24639382
- [Background] Wanders LK, East JE, Uitentuis SE, Leeflang MM, Dekker E. Diagnostic performance of narrowed spectrum endoscopy, autofluorescence imaging, and confocal laser endomicroscopy for optical diagnosis of colonic polyps: a meta-analysis. Lancet Oncol. 2013 Dec;14(13):1337-47. doi: 10.1016/S1470-2045(13)70509-6. Epub 2013 Nov 13. PMID 24239209
- [Background] Kaltenbach T, Rex DK, Wilson A, Hewett DG, Sanduleanu S, Rastogi A, Wallace M, Soetikno R. Implementation of optical diagnosis for colorectal polyps: standardization of studies is needed. Clin Gastroenterol Hepatol. 2015 Jan;13(1):6-10.e1. doi: 10.1016/j.cgh.2014.10.009. No abstract available. PMID 25511846
- [Background] Kumar S, Fioritto A, Mitani A, Desai M, Gunaratnam N, Ladabaum U. Optical biopsy of sessile serrated adenomas: do these lesions resemble hyperplastic polyps under narrow-band imaging? Gastrointest Endosc. 2013 Dec;78(6):902-909. doi: 10.1016/j.gie.2013.06.004. Epub 2013 Jul 9. PMID 23849819
- [Background] Hazewinkel Y, Lopez-Ceron M, East JE, Rastogi A, Pellise M, Nakajima T, van Eeden S, Tytgat KM, Fockens P, Dekker E. Endoscopic features of sessile serrated adenomas: validation by international experts using high-resolution white-light endoscopy and narrow-band imaging. Gastrointest Endosc. 2013 Jun;77(6):916-24. doi: 10.1016/j.gie.2012.12.018. Epub 2013 Feb 21. PMID 23433877
- [Derived] Vleugels JLA, Hazewinkel Y, Dijkgraaf MGW, Koens L, Fockens P, Dekker E; DISCOUNT study group. Optical diagnosis expanded to small polyps: post-hoc analysis of diagnostic performance in a prospective multicenter study. Endoscopy. 2019 Mar;51(3):244-252. doi: 10.1055/a-0759-1605. Epub 2018 Dec 13. PMID 30544284